CLINICAL TRIAL: NCT00891579
Title: Phase 2 Randomized, Controlled, Open-label Study of Pemetrexed Versus Gefitinib in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer Who Have Previously Received Platinum-Based Chemotherapy Without EGFR Mutations
Brief Title: Study of Pemetrexed Versus Gefitinib in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer Who Have Previously Received Platinum-Based Chemotherapy Without Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Director of Chinese Society of Lung Cancer/Chief of Lung Cancer Research Institute & Cancer Center/Vice President of Guangdong General hospital, Chinese Society of Lung Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG0806
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; EGFR; Pemetrexed; Gefitinib; without EGFR mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gefitinib

ARMS (2):
- Alimta (Active Comparator): Treatment of Alimta
  Interventions: Drug: Pemetrexed (Alimta)
- IRESSA (Active Comparator): Treatment of IRESSA
  Interventions: Drug: Gefitinib (IRESSA)

INTERVENTIONS:
Drug: Pemetrexed (Alimta) — treatment of single pemetrexed with vitamin supplement until discontinued conditions are met
  Arms: Alimta
Drug: Gefitinib (IRESSA) — treatment of Gefitinib will be applied until discontinued conditions are met
  Arms: IRESSA

SUMMARY:
This study is a prospective trial of Alimta (pemetrexed) versus IRESSA (gefitinib) among epidermal growth factor receptor wild-type Non-Small Cell Lung Cancer (NSCLC) patients in a 2nd line setting.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be signed.
2. At least 18 years of age.
3. Histologic or cytologic diagnosis of NSCLC.
4. Locally advanced or metastatic disease (stage IIIB, or IV) that is not amenable to definitive surgery or radiotherapy.
5. Patients must have previously received one platinum-based chemotherapy regimen for palliative therapy of locally advanced or metastatic disease. Patients are also eligible if they have received one platinum-based chemotherapy regimen as neoadjuvant or adjuvant chemotherapy and the disease recurred within six months since the finishing of neoadjuvant or adjuvant chemotherapy.
6. Without EGFR mutations.
7. At least one measurable lesion as defined by RECIST criteria.
8. ECOG PS0 - 2.
9. Adequate organ function including the following:

   * bone marrow;
   * hepatic;
   * renal.
10. Prior chemotherapy must be completed at least 3 weeks prior to the study enrollment, and the patient must have recovered from the toxic effects of the treatment (except for alopecia).
11. Previous palliative radiation therapy is allowed, but limited in LESS 25% of the bone marrow and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed one month before study entry. Radiotherapy should not be administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented.
12. Estimated life expectancy of at least 8 weeks.
13. For women:

    * must be surgically sterile;
    * postmenopausal; OR
    * compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period; must have negative serum or urine pregnancy test and must not be lactating.
14. For men:

    * must be surgically sterile; OR
    * compliant with a contraceptive regimen during and for 3 months after the treatment period.
15. Patient compliance and geographic proximity that allow adequate follow-up.

Exclusion Criteria:

1. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry or concurrent administration of any other anti-tumor therapy.
2. Have previously participated in a study involving pemetrexed or EGFR-TKI
3. Hypersensitivity to pemetrexed or gefitinib or any ingredients in the two drugs.
4. Symptomatic central nervous system (CNS) metastases and asymptomatic CNS metastases requiring concurrent corticosteroid therapy. Treated stable CNS metastases are allowed; the patient must be stable after radiotherapy for more than 2 weeks and off of corticosteroids for more than 1 week. .
5. History of another malignancy within the last 5 years except cured carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and superficial bladder tumors (Ta, Tis and T1)
6. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
7. Patients with interstitial lung disease.
8. Any unstable systemic disease (including active infection, hepatic, renal or metabolic disease) or serious concomitant disorders that would compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
9. Significant cardiovascular event: congestive heart failure >NYHA class 2; unstable angina, active CAD (myocardial infarction more than 1 year prior to study entry is allowed); serious cardiac arrhythmia requiring antiarrythmic therapy ( beta blockers or digoxin are permitted) or uncontrolled hypertension.
10. History of significant neurological or mental disorder, including seizures or dementia.
11. Incision from operation has not healed before the start of study treatment (Small incision for biopsy is eligible.)
12. Pregnant or breast-feeding women and childbearing potential women with either a positive or no pregnancy test within 48 hours of the start of treatment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.
13. Concurrent use of St. John's Wort, Rifampicin, and/or ritonavir.
14. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed. If a patient is taking an NSAID (Cox-2 inhibitors included) or salicylate with a long half-life (e.g., naproxen, piroxicam, diflunisal, nabumetone, rofecoxib, or celecoxib) it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed.
15. Presence of clinically detectable (by physical exam) third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
16. Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2009-02; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years

SECONDARY OUTCOMES:
Response rate (RR) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Lung Cancer Research Institute & Cancer Center of Guangdong General Hospital, Guangzhou, Guangdong
  - 307 hospital of People's Liberation Army, Beijing
  - Peking Union Hospital, Beijing
  - Jilin Tumor Hospital, Changchun
  - Nanjing General Hospital of Nanjing Military Command, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - The first hospital of China medical university, Shenyang

REFERENCES:
- [Derived] Zhou Q, Cheng Y, Yang JJ, Zhao MF, Zhang L, Zhang XC, Chen ZH, Yan HH, Song Y, Chen JH, Feng WN, Xu CR, Wang Z, Chen HJ, Zhong WZ, Liu YP, Wu YL. Pemetrexed versus gefitinib as a second-line treatment in advanced nonsquamous nonsmall-cell lung cancer patients harboring wild-type EGFR (CTONG0806): a multicenter randomized trial. Ann Oncol. 2014 Dec;25(12):2385-2391. doi: 10.1093/annonc/mdu463. Epub 2014 Oct 3. PMID 25281710